CLINICAL TRIAL: NCT02599363
Title: A Phase I Trial of Ribocilcib (LEE011) and Weekly Paclitaxel in Patients With Rb+ Advanced Breast Cancer
Brief Title: A Trial of Ribocilcib (LEE011) and Weekly Paclitaxel in Patients With Rb+ Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 06115
Record Dates: First submitted 2015-11-05; First posted 2015-11-06 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — ribociclib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Escalation Treatment Arm (Experimental)
  Interventions: Drug: Ribociclib (LEE011); Drug: Paclitaxel

INTERVENTIONS:
Drug: Ribociclib (LEE011)
Drug: Paclitaxel

SUMMARY:
This is a Phase I study to assess the safety and Maximum tolerated dose (MTD) of paclitaxel + ribociclib (LEE011) in patients with Rb+, advanced breast cancer. Dose escalation will be performed using standard 3 + 3 dosing strategy. The starting dose of ribociclib (LEE011) is 200 mg once daily; dose escalation proceeds in 200 mg increments up to a maximum of 600 mg. Dose-limiting toxicities (DLT) will be based upon first-cycle toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or cytologically confirmed breast cancer that is now metastatic; any ER, PR or HER2 status is allowed.
* Biopsy confirming metastatic breast cancer and Retinoblastoma protein (Rb) positivity by immunohistochemistry prior to enrolling on this protocol is required.
* Biopsy must be obtained immediately before study enrollment; no intervening treatments are allowed.
* Patient must have measurable disease defined by RECIST 1.1 criteria.
* Age ≥18 years
* Patient must have received ≤3 prior cytotoxic regimens in the metastatic setting.
* Performance status of 0-1 on the ECOG Performance Scale.
* The subject must have adequate organ function, defined as follows

  * Serum creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 50 mL/min
  * In the absence of liver metastases, alanine aminotransferase (AST) and aspartate aminotransferase (ALT) < 2.5 x ULN. If the patient has liver metastases, ALT and AST < 5 x ULN.
  * Total bilirubin < ULN; or total bilirubin ≤ 3.0 x ULN or direct bilirubin ≤ 1.5 x ULN in patients with well documented Gilbert's Syndrome.
  * For subjects without extensive bone metastases: alkaline phosphatase levels < 2.5 x ULN
  * Potassium, total calcium (corrected for serum albumin), magnesium, sodium and phosphorus within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication
  * INR ≤ 1.5 unless on warfarin in which case INR <3.0 is acceptable.
* The subject must have adequate marrow function, defined as follows

  * Leukocytes Absolute neutrophil count (ANC) ≥1500/mm3
  * Platelets ≥100,000/mm3, and
  * Hemoglobin ≥9 g/dL
* The subject must be able to swallow ribociclib (LEE011)

Exclusion Criteria

* Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of Study Day 1 or within 5 half-lives of the investigational product, whichever is longer, with the exception of a prior CDK 4/6 inhibitor.
* Patient has had prior toxicity from a CDK 4/6 inhibitor necessitating discontinuation of the drug. Patient may have had prior treatment with a cdk 4/6 inhibitor in the adjuvant or metastatic setting.
* Patient who has had chemotherapy or exposure to a CDK 4/6 inhibitor within 3 weeks (6 weeks for nitrosoureas, mitomycin C or bevacizumab) who has not recovered from the adverse events due to previous agents administered more than 4 weeks prior to Study Day 1. Hormonal therapy must be discontinued at least 24 hours prior to starting study treatment.
* Patient is unable to have a biopsy of a metastatic site for Rb testing, because the biopsy is felt to be too invasive or risky by the treating physician.
* Patient has not received available therapies that confer clinical benefit.
* Patient has known active CNS metastases and/or carcinomatous meningitis. However, patients with CNS metastases (including brain metastases) are eligible for the study provided they are clinically stable and have met ALL of the following criteria:
* At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment
* Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases.
* Patient has known hypersensitivity to any of the excipients of ribociclib
* The subject has uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Diabetes mellitus
  * Symptomatic congestive heart failure (see 5.2.14), unstable angina pectoris, stroke or myocardial infarction within 12 months of screening
* Patient has baseline neuropathy of ≥ grade 2.
* Patients who have known allergic reactions to paclitaxel or IV contrast dye despite standard prophylaxis.
* The subject is known to be positive for the human immunodeficiency virus (HIV). Note: baseline HIV screening is not required
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.
* Patient has a concurrent malignancy or malignancy within 3 years prior to starting study drug, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer.
* Patient is not able to swallow oral medication and/or has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.).
* Patient has active cardiac disease or a history of cardiac dysfunction including any of the following:
* History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 12 months prior to screening
* History of documented congestive heart failure (New York Heart Association functional classification III-IV)
* Documented cardiomyopathy
* Patient has a Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) at screening
* History of ventricular, supraventricular, nodal arrhythmias, or any other cardiac arrhythmias, long QT Syndrome or conduction abnormality within 12 months of screening
* Congenital long QT syndrome or family history of long QT syndrome
* Bradycardia (heart rate <50 at rest), by ECG or pulse, at screening
* Systolic blood pressure (SBP) > 160 mmHg or < 90 mmHg at screening
* On screening, inability to determine the QTcF interval on the ECG (i.e.: unreadable or not interpretable) or QTcF > 450 msec (using Fridericia's correction). All as determined by screening ECG (mean of triplicate ECGs)
* Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to starting study drug (see Table 6.2 for details):
* Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pummelos, star-fruit, and Seville oranges
* That have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
* That have a known risk to prolong the QT interval or induce Torsades de Pointes
* Patient is currently receiving or has received systemic corticosteroids ≤ 2 weeks prior to starting study drug, or has not fully recovered from side effects of such treatment. The following uses of corticosteroids are permitted: single doses, topical application (e.g., for rash), inhaled sprays (e.g., for obstructive airway diseases), eye drops or local injections (e.g., intra-articular).
* Patient is currently receiving warfarin or other coumarin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed.
* Participation in a prior investigational therapeutic study within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer.
* Patient who has received radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug, and who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia) and/or in whom ≥ 25% of the bone marrow was irradiated.
* Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (all surgical wounds must be fully healed). For the purpose of this criterion, a major surgical procedure is defined as one requiring the administration of general anesthesia (tumor biopsy is not considered as major surgery).
* Patient has not recovered from all toxicities related to prior anticancer therapies to NCI-CTCAE version 4.03 Grade <1 (Exception to this criterion: patients with any degree of alopecia are allowed to enter the study).
* Patient with a Child-Pugh score B or C
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception throughout the study and for 8 weeks after study drug discontinuation. Highly effective contraception methods include:
* Total abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
* Combination of any two of the following (a+b or a+c or b+c) Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception Placement of an intrauterine device (IUD) or intrauterine system (IUS) Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository
* In case of use of oral contraception, women should have been stable on the same pill before taking study treatment.
* Note: Oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction.
* Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01; Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Amy Clark, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States